CLINICAL TRIAL: NCT01423240
Title: A Randomized, 6-week, Double-blind, Placebo-controlled, Fixed-dose, Parallel Group Study of Lurasidone for the Treatment of Major Depressive Disorder With Mixed Features
Brief Title: Major Depressive Disorder With Mixed Features
Acronym: RESOLVE2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050305
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Lurasidone; Latuda
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone 20 mg (Experimental)
  Interventions: Drug: Lurasidone 20 mg
- Lurasidone 60 mg (Experimental)
  Interventions: Drug: Lurasidone 60 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone 20 mg — Lurasidone 20 mg once daily orally in the evening
  Other Names: Latuda
  Arms: Lurasidone 20 mg
Drug: Lurasidone 60 mg — Lurasidone 60 mg once daily orally in the evening
  Other Names: Latuda
  Arms: Lurasidone 60 mg
Drug: Placebo — Placebo once daily orally in the evening
  Arms: Placebo

SUMMARY:
Lurasidone HCl is a compound that is a candidate for the treatment of major depressive with mixed features.This clinical study is designed to test how well Lurasidone works to treat major depressive disorder with mixed features.

ELIGIBILITY:
Inclusion Criteria:

Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.

Subject is 18 to 75 years of age, inclusive. Subject has MDD (diagnosed by DSM-IV-TR, and confirmed by the Structured Clinical Interview for DSM-IV Disorders - Clinical Trial version [SCID-CT]).

Subject is currently experiencing a major depressive episode (diagnosed by DSM-IV-TR; at least 2 weeks in duration) AND two or three of the following manic symptoms occurring on most days over at least the last 2 weeks (confirmed by the SCID-CT modified for Study D1050305):

* Elevated, expansive mood
* Inflated self-esteem or grandiosity
* More talkative than usual or pressure to keep talking
* Flight of ideas or subjective experience that thoughts are racing
* Increase in energy or goal-directed activity (either socially, at work or school, or sexually)
* Increased or excessive involvement in activities that have a high potential for painful consequences (e.g., engaging in unrestrained buying sprees, sexual indiscretions, or foolish business investments)
* Decreased need for sleep (feeling rested despite sleeping less than usual; to be contrasted from insomnia) Subject has a rater-administered Montgomery-Asberg Depression Rating Scale (MADRS) total score of ≥ 26 at screening and both a rater-administered and self-rated (administered by computer) MADRS total score ≥ 26 at baseline.

Exclusion Criteria:

Subject has Axis I or Axis II diagnosis other than MDD that has been the primary focus of treatment within the 3 months prior to screening Subject answers "yes" to "Suicidal Ideation" Item 4 or 5 on the C-SSRS (at time of evaluation) at screening or baseline visit.

Subject has attempted suicide within the past 3 months. Subject has a lifetime history of any bipolar I manic or mixed manic episode. Subject has any abnormal laboratory parameter at screening that indicates a clinically significant medical condition as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
MADRS | 6 weeks
  Mean change from baseline in MADRS total score after 6 weeks of treatment

SECONDARY OUTCOMES:
CGI-S | 6 weeks
  Global severity assessed by the CGI-S score (depression)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (27):
- United States (27):
  - Birmingham Research Group, Birmingham, Alabama
  - Sun Valley Behavioral Medical, Imperial, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Pacific Clinical Research Medical Group, Orange, California
  - SMRI, Sherman Oaks, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Florida Research Center, Maitland, Florida
  - University of Miami, Miller School, Miami, Florida
  - Miami Research, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive NeuroScience Inc., Atlanta, Georgia
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Psychiatric Medicine Associates, Skokie, Illinois
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - CRI Worldwide, Willingboro, New Jersey
  - Medical & Behavioral Health Research, New York, New York
  - Montefiore Medical Center; Anxiety & Depression Clinic; Dept. of Psychiatry, The Bronx, New York
  - New Hope Clinical Research, Hickory, North Carolina
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Harry Croft and Associates, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Department of Psychiatry, University of Utah Health Sciences Center, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Derived] Goldberg JF, Siu C, Mao Y, Tsai J, Pikalov A, Calabrese JR, Loebel A. Major depressive disorder with mixed features and treatment response to lurasidone: A symptom network model. J Affect Disord. 2020 Dec 1;277:1045-1054. doi: 10.1016/j.jad.2020.08.048. Epub 2020 Aug 26. PMID 33065813
- [Derived] Suppes T, Silva R, Cucchiaro J, Mao Y, Targum S, Streicher C, Pikalov A, Loebel A. Lurasidone for the Treatment of Major Depressive Disorder With Mixed Features: A Randomized, Double-Blind, Placebo-Controlled Study. Am J Psychiatry. 2016 Apr 1;173(4):400-7. doi: 10.1176/appi.ajp.2015.15060770. Epub 2015 Nov 10. PMID 26552942